CLINICAL TRIAL: NCT00750659
Title: Open-label Trial of Nilotinib in Patients With Advanced (>CP1) Chronic Myeloid Leukemia or Ph+ Acute Lymphatic Leukemia Pre- and Post- Allogeneic Stem Cell Transplantation.
Brief Title: Nilotinib Pre and Post Allogeneic Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-08-5288-AN-CTIL
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Chronic Myeloid Leukemia; Acute Lymphoblastic Leukemia; Stem Cell Transplantation
Keywords: Chronic myeloid leukemia; Ph+ acute lymphoblastic leukemia; stem cell transplantation; nilotinib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Nilotinib treatment
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib — Nilotinib 400 mg po/BID until transplant. Nilotinib 200-400 mg po/BID post transplant in escalated doses.

SUMMARY:
Current therapeutic results in advanced chronic myeloid leukemia (CML) and Ph+ acute lymphoblastic leukemia (ALL) are rather disappointing. Most of these patients will eventually undergo allogeneic stem cell transplantation. Nilotinib is a novel TKI tyrosine kinase inhibitor with 30 fold more potency than Imatinib. Based on previous preliminary experience the author we rationalize that Nilotinib therapy pre- allogeneic transplantation for patients with advanced CML and Ph+ALL will reduce tumor mass pre- transplant achieving a state of minimal residual disease (MRD) and therefore may improve transplantation outcome without increasing toxicity. In addition it will allow time for improving patient medical condition and for finding an unrelated donor which will enable allogeneic transplantation , and to induce anti tumor effect post PBSC w\o DLI ( donor lymphocyte infusion)

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Ph+ advanced CML (>CR1) or Ph+ALL.
2. Hematological, Cytogenetic (Ph+) and/or BCR/ABL positive documented at diagnosis of CML or Ph+ALL pre- alloSCT.
3. Patients age 18-65 years of age.
4. .Patients must have an HLA compatible donor willing and capable of donating peripheral blood stem cells (first choice) or bone marrow progenitor cells using conventional techniques, and blood lymphocytes if indicated (HLA compatible defined as 5/6 or 6/6 matched related or matched unrelated donor.
5. Adequate end organ function, defined as the following:

   total bilirubin < 1.5 x ULN, SGOT and SGPT < 2.5 x UNL , creatinine < 1.5 x ULN
6. Patient must have LVEF>45% prior entry into study.
7. Patient must have QTc <450 msec at study entry.
8. Lung diffusion capacity (DLCO>40% predicted)
9. Female patients of childbearing potential must have negative pregnancy test within 7 days before initiation of study drug dosing. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Male and female patients of reproductive potential must agree to employ an effective barrier method of birth control throughout the study and for up to 3 months following discontinuation of study drug.
10. Written, voluntary informed consent.

Exclusion Criteria:

1. Patients with CML in first chronic phase
2. Patient has received any other investigational agents within 28 days of first day of study drug dosing, unless the disease is rapidly progressing.
3. ECOG performance status > 2
4. Patient is < 5 years free of another primary malignancy except: if the other primary malignancy is not currently clinically significant nor requiring active intervention, or if other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ. Existence of any other malignant disease is not allowed.
5. Impaired cardiac function including any one of the following:

   * LVEF < 45% or below the institutional lower limit of the normal range (whichever is higher) as determined by echocardiogram
   * Inability to determine the QT interval on ECG
   * Complete left bundle branch block
   * Long QT syndrome or a known family history of long QT syndrome.
   * Clinically significant resting bradycardia (<50 beats per minute)
   * QTc > 450 msec on baseline ECG (using the QTcF formula). If QTcF >450 msec and electrolytes are not within normal ranges, electrolytes should be corrected and then the patient re-screened for QTc
   * Myocardial infarction within 12 months prior to starting study
   * Other clinically significant heart disease (e.g. unstable angina, congestive heart failure or uncontrolled hypertension).
6. Female patients who are pregnant or breast-feeding.
7. Patient has a severe and/or uncontrolled medical disease (i.e., uncontrolled diabetes, chronic renal disease, or active uncontrolled infection).
8. Patient has known chronic liver disease (i.e., chronic active hepatitis, and cirrhosis).
9. Patient has a known diagnosis of human immunodeficiency virus (HIV) infection.
10. Patient had a major surgery within 2 weeks prior to study entry.
11. Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.
12. Patients with active CNS disease (patients with history of CNS disease are allowed).
13. Patients with pleural effusion or ascites
14. Patients with a history of pancreatitis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Safety | 12 months

SECONDARY OUTCOMES:
response | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Nagler, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Chaim Sheba Medical Center, Tel Litwinsky, Israel

REFERENCES:
- [Derived] Shimoni A, Volchek Y, Koren-Michowitz M, Varda-Bloom N, Somech R, Shem-Tov N, Yerushalmi R, Nagler A. Phase 1/2 study of nilotinib prophylaxis after allogeneic stem cell transplantation in patients with advanced chronic myeloid leukemia or Philadelphia chromosome-positive acute lymphoblastic leukemia. Cancer. 2015 Mar 15;121(6):863-71. doi: 10.1002/cncr.29141. Epub 2014 Nov 11. PMID 25387866